CLINICAL TRIAL: NCT03649438
Title: 131I-Metaiodobenzylguanidine (131I-MIBG) Therapy for Relapsed/Refractory Neuroblastoma
Status: No longer available | Type: Expanded Access
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Tanya Watt, Assistant Professor, University of Texas Southwestern Medical Center
Other Study IDs: STU-2019-0665
Record Dates: First submitted 2018-07-18; First posted 2018-08-28 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Relapsed Neuroblastoma; Metastatic Pheochromocytoma
MeSH Terms: conditions — Neuroblastoma; Pheochromocytoma | interventions — 3-Iodobenzylguanidine; Potassium Iodide; Granulocyte Colony-Stimulating Factor; pegfilgrastim

STUDY DESIGN:
Expanded Access Types: Intermediate, Treatment

INTERVENTIONS:
Drug: 131 I-Metaiodobenzylguanidine — * Minimum dose of 10 mCi/kg for patients without a stem cell source whose renal function is above the upper limit of normal but still meets eligibility criteria.
  * Dose of 12 mCi/kg for patients without a stem cell source with normal renal function and meets other eligibility criteria.
  * Dose of > 12 mCi/kg to 18 mCi/kg maximum at investigator's discretion for patients meeting eligibility criteria with stem cells available.
  Other Names: 131I-MIBG
Drug: Potassium Iodide — For the therapeutic MIBG administration, potassium iodide solution will be administered in a loading dose of 6mg/kg orally at least 8 hours prior to the MIBG injection, and then will be given at 1mg/kg/dose every 4 hours on days 0-6, then 1 mg/kg/day through day 45 post injection.
  Other Names: KI solution
Drug: G-csf — It is recommended that patients with ANC less than 750 after MIBG infusion begin G-CSF 5 mcg/kg/day subcutaneously (or receive equivalent single dose of Neulasta every 14 days while neutropenic) until neutrophil recovery (generally >5000). This will start 24 hours after stem cell infusion (if stem cells are to be infused).
  Other Names: Neulasta

SUMMARY:
This expanded access is the best available therapy/compassionate use designed to determine the palliative benefit and toxicity of 131I-MIBG in patients with relapsed/refractory neuroblastoma or metastatic pheochromocytoma who are not eligible for therapies of higher priority. Patients may receive a range of doses depending on stem cell availability and tumor involvement of bone marrow. Response rate, toxicity, and time to progression and death will be evaluated.

DETAILED DESCRIPTION:
Primary Objective is to provide access to therapy with 131I-MIBG for patients with relapsed/refractory neuroblastoma or metastatic pheochromocytoma.

Secondary Objectives are to (1) assess disease response to 131I-MIBG therapy for patients with relapsed/refractory neuroblastoma or metastatic pheochromocytoma; (2) gain more information about the toxicities of 131I-MIBG therapy; and (3) assess improvement of symptoms, including pain and fatigue, for patients with relapsed/refractory neuroblastoma or metastatic pheochromocytoma who are receiving 131I-MIBG therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis:
* Relapsed/refractory neuroblastoma with original diagnosis based on tumor histopathology or elevated urine catecholamines with typical neuroblastoma cells in the bone marrow
* Metastatic pheochromocytoma
* Age >1 year and able to cooperate with radiation safety restrictions during therapy period
* Karnofsky or Lansky performance status of ≥ 50%
* Life expectancy: patients must have a life expectancy of at least 8 weeks
* Disease status: Failure to respond to standard therapy (usually combination chemotherapy with or without radiation and surgery) or development of progressive disease at any phase of standard therapy (any new lesion or an increase in size >25% of a pre-existing lesion). Patients may enter this study with or without re-induction therapy for recurrent tumor.
* Disease must be evaluable by MIBG scan. A positive MIBG scan must be present within 8 weeks prior to study entry and subsequent to any intervening therapy. If the patient has only one MIBG positive lesion and that lesion was radiated, a biopsy must be done at least 4 weeks after radiation was completed and must show viable neuroblastoma.
* Stem Cells: If a patient does not have a hematopoietic stem cell product available for re-infusion after MIBG treatment, they may not receive a 131IMIBG dose >12 mCi/kg. Patients must have a hematopoietic stem cell product available for re-infusion after MIBG treatment at doses of > 12 mCi/kg. The minimum quantity for peripheral blood stem cells is 1.5 x 106 CD34+ cells/kg (optimum > 2 x 106 CD34+ cells/kg). The minimum dose for bone marrow is 1.0 x 108 mononuclear cells/kg (optimum >2.0 x 108 mononuclear cells/kg).
* Stem cell source: The patients on this protocol will have autologous PBSCs available.
* Have acceptable organ function as defined below within 7 days of enrollment:
* Bone Marrow: ANC ≥750 X 109 /L, platelets ≥50,000 X 109 /L, and hemoglobin ≥ 8.0 g/dL without transfusion if stem cells are not available. ANC ≥500 X 109 /L, platelets ≥20,000 X 109 /L, and hemoglobin ≥ 8.0 g/dL with transfusions allowed if stem cells are available. Patients with stem cells available are excluded if they require two platelet transfusions per week to maintain the minimum required platelet count. A bone marrow examination is not medically indicated for patients diagnosed with metastatic pheochromocytoma.
* Renal: Creatinine ≤ 2 times upper limit of normal
* Hepatic: Bilirubin ≤2x upper limit of normal; AST/ALT ≤10x upper limit of normal
* Cardiac: Ejection fraction ≥ 45% on echocardiogram or shortening fraction

  >/=27%
* Pulmonary: normal lung function as manifested by no dyspnea and/or oxygen saturation ≥ 94% on room air.
* Prior Therapy: Patients must have recovered from all acute toxicities (defined as CTCAE 5.0 ≤ grade 1) associated with any prior therapy, and:
* Myelosuppressive chemotherapy: At least 2 weeks should have elapsed since any chemotherapy causing myelosuppression
* Biologic (anti-neoplastic agent): At least 7 days should have elapsed since the completion of therapy with a biologic agent.
* Monoclonal antibodies: At least 3 half-lives should have elapsed since therapy with a monoclonal antibody
* Radiation therapy: Three-months should have elapsed in the case of completing radiation to any of the following fields: craniospinal, total abdominal, whole lung, total body irradiation). For all other sites of radiation, at least 2 weeks should have elapsed.
* Cytokine therapy (e.g. G-CSF, GM-CSF, IL-6, IL-2): must be discontinued a minimum of 24 hours prior to MIBG therapy.
* Voluntary written informed consent must be obtained before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.

Exclusion Criteria:

* Patients with disease of any major organ system that would compromise their ability to withstand therapy.
* Because of the teratogenic potential of the study medication, no patients who are pregnant or lactating will be allowed. Patients of childbearing potential must practice an effective method of birth control while participating on this study, to avoid possible damage to the fetus.
* Known allergy to any of the agents or their ingredients used in this study.
* Patients who are on hemodialysis
* Patients with untreated positive blood cultures or progressive infections as assessed by radiographic studies
* Patients who have had prior treatment with 131I-MIBG who do not meet the re-treatment criteria.
* In patients with metastatic pheochromocytoma, screening urinalysis required prior to study enrollment. If random collection urine specimen is positive for proteinuria, patients must have 24-hour urine protein determination. Patients with metastatic pheochromocytoma are excluded if 24-hour urine protein is above the institutional upper limit of normal.
* Patients with known MIBG-avid parenchymal brain metastases are excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Watt, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- The University of Texas Southwestern Medical Center, Dallas, Texas, United States